CLINICAL TRIAL: NCT04939753
Title: Incidence of Nephrogenic Diabetes Insipidus During Prolonged Sevoflurane Sedation in the Intensive Care Unit: a Retrospective Analysis
Brief Title: Nephrogenic Diabetes Insipidus During Prolonged Sevoflurane Sedation in the ICU: a Retrospective Analysis
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: Sevoflu-DI-IZ
Record Dates: First submitted 2021-04-27; First posted 2021-06-25 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Nephrogenic Diabetes Insipidus
MeSH Terms: conditions — Diabetes Insipidus, Nephrogenic | interventions — Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sevoflurane group: Patients that received sevoflurane while in ICU care.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane administration to sedate the patient

SUMMARY:
The investigators aim to retrospectively explore the electronic medical records of all patients who were admitted to the Intensive Care Unit (ICU) of the UZ Brussels in the last 10 years (March 1st 2011- March 1st 2021) and who received prolonged sedation (>24h) with sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* Sevoflurane administration >24h
* 18 years and older

Exclusion Criteria:

* < 18 years old
* Pre-existing diabetes insipidus
* Use of drugs at risk for diabetes insipidus (including lithium, cisplatin)
* Hypercalcemia (persistently >2.75 mmol/L)
* Pituitary or acute brain surgery
* Patients requiring continuous renal replacement therapy
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all patients who were admitted to the Intensive Care Unit (ICU) of the UZ Brussels in the last 10 years (March 1st 2011- March 1st 2021) and who received prolonged sedation (>24h) with sevoflurane.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Nephrogenic Diabetes Insipidus prevalence | up to 8 weeks
  How many patients under sevoflurane sedation ultimately develop NDI? NDI confirmed by demonstrating the absence of a urine concentrating response to exogenous Arginine Vasopressine.

SECONDARY OUTCOMES:
Number of patients that develop risk factors of NDI | up to 8 weeks
  Number of patients that develop risk factors (electrolyte disorder, urinary obstruction) for NDI.
Amount of time patient was placed under sevoflurane sedation. | up to 8 weeks
  How long are they under sevoflurane sedation.
Number of patients with electrolyte abnormalities as assessed by lab results. | during hospitalization, up to 8 weeks.
  Lab results of hematology and chemistry labs show an electrolyte imbalance.
Number of patients with excessive urine output | during hospitalization, up to 8 weeks.
  Amount of urine output: >40 ml/kg/24h
Number of patients with an abnormal physical examination. | during hospitalization, up to 8 weeks.
  Typical physical symptoms of (N)DI: tired, lethargic, tachycardia, tachypnea, hypotension and dry mucous membranes.
Number of patients with urine with an abnormal osmolality | during hospitalization, up to 8 weeks.
  Lab testing of urine: osmolality < 300 mosm/kg
Number of patients that show an abnormal amount of fluid intake | during hospitalization, up to 8 weeks.
  >2.5l/day
Number of patients that have an abnormal abdominal echo of the bladder. | during hospitalization, up to 8 weeks.
  Echo shows an enlarged bladder.
Number of symptoms of NDI | up to 8 weeks
  Number of symptoms of NDI do these patients show?
Timing of symptoms of NDI | up to 8 weeks
  After how much time do these patients show symptoms of NDI?

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided